CLINICAL TRIAL: NCT02082613
Title: Lord´s Procedure Versus Sclerotherapy for Testicular Hydrocele; a Randomized Controlled Study.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Karl-Johan Lundström, MD, resident Urologist, Umeå University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JLL-378961
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Testicular Hydrocele
Keywords: Testicular hydrocele; Hydrocele; Sclerotherapy; Surgery; Complications
MeSH Terms: conditions — Testicular Hydrocele | interventions — Sclerotherapy; Polidocanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lord´s procedure (Experimental): Lord´s procedure for testicular hydrocele, under local anesthesia in a conventional operation room, under sterile conditions
  Interventions: Procedure: Lord´s procedure
- Sclerotherapy (Active Comparator): Sclerotherapy with 4 ml of polidocanol 30mg/ml after complete emptying of the hydrocele. With or without local anesthesia, not performed in an operation room.
  Interventions: Procedure: Sclerotherapy

INTERVENTIONS:
Procedure: Lord´s procedure
  Arms: Lord´s procedure
Procedure: Sclerotherapy
  Other Names: Polidocanol 30mg/ml, 4ml; Aetoxysclerol™ 30mg/ml, 4ml; Lauromakrogol 400 30mg/ml, 4ml
  Arms: Sclerotherapy

SUMMARY:
This study will compare a minimal invasive operation in local anesthesia with sclerotherapy for symptomatic testicular hydrocele within 6 months after randomization. Thirty days complication rates will be assessed. The hypothesis is that surgery will lead to faster cure while sclerotherapy would be cheaper and have less complications.

DETAILED DESCRIPTION:
Testicular hydrocele is a common disorder even though it´s exact prevalence is unknown. In areas with filariasis it´s endemic.

Hydrocele is a benign condition where fluid accumulates in between two layers of tunica vaginalis (embryologically, the peritoneum), surrounding the testicle. The cause is unknown but inflammatory conditions is believed to induce these changes. The pathogenesis of hydrocele is believed to be a nonbalanced secretion and resorption of fluid.

Diagnosis of hydrocele is easy since the patient presents with an enlarged scrotum and clinical investigation including palpation and transillumination of the scrotum confirms the diagnosis. A scrotal ultrasound might be indicated to rule out a malignancy or if the diagnosis is unclear.

Treatment for hydrocele is only indicated when the patient has symptoms since all treatment modalities carries risk of complications, such as hematoma, infection, pain and even infertility concerns has been raised.

Operative management is considered the golden standard of treatment when considering recurrence but less invasive procedures such as sclerotherapy is frequently used, mainly due to cost and complications issues.

Lord´s procedure has in several series shown low frequency of complications and excellent recurrence rates. However, Lord´s procedure and sclerotherapy has not been tested head to head and the optimal treatment for hydrocele is yet to be determined.

This study aims to compare these techniques and evaluate the results within 1 year after randomization on cure, complication rates and various secondary descriptive outcomes.

The investigators aim to adhere to CONSORT.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic testicular hydrocele, with more than 2 points on a validated inguinal botherscore (Inguinal Pain Questionnaire, IPQ)
* More than 40ml of hydrocele fluid
* Age>40 years
* Completed reproduction
* Oral and written consent to participate in the study
* American Association of Anesthesiology (ASA) grade≤ 3

Exclusion Criteria:

* Other ipsilateral scrotal disease (tumour, ongoing inflammatory disease of the scrotum,)
* Ongoing urinary infection
* Ipsilateral inguinal hernia
* Ascites
* Paternity wish
* Not possible to drain the hydrocele fully
* Opaque fluid drained on emptying the hydrocele
* Bilateral hydrocele where both sides has symptom score more than 2p on IPQ.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-12 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Cure from symptomatic hydrocele within 6 months of randomization | Every 3 months until 6months from randomization

SECONDARY OUTCOMES:
Postoperative complications | Within 30 days from treatment

OTHER OUTCOMES:
Proportion symptomatic scrotal complaints without recurrence of hydrocele | 6 months
Proportion treatment failure | 6 months
  The proportion of men who in this combined outcome showed either recurrence, significant symptoms but refuses further treatment, residual symptoms without hydrocele or patient preference to change treatment modality, converting from one treatment arm to the other.
Mean number of treatments until cure | 6 months
Mean days on sick leave | 30 days
Proportion cured by solely emptying the hydrocele | 2-3months
  Patients who are randomized to surgery will undergo an emptying of the hydrocele to allow for clinical examination of the testicle. The amount will be measured and inspected. No sclerotherapy will be instilled. If patients are cured by this simple measure, they will be classified as cured by this and analyzed as cured by surgery, in intention to treat analysis.
Description of inconvenience grade of patients with hydrocele | First visit
  The inconvenience grade for patients presenting in a urological out patient setting, reported as a 7 scale question, (adopted from Inguinal Pain questionnaire).

CONTACTS AND LOCATIONS:
Overall Officials: Pär Nordin, Ph.D, MD, Study Director — Umeå University; Karl-Johan Lundström, M.D, Principal Investigator — Östersunds Hospital
Locations (7):
- Drammen Hospital, Drammen, Norway
- Sweden (6):
  - Falu lasarett, Falun, Dalarna County
  - Östersunds hospital, Östersund, Jämtland County
  - Helsingborgs sjukhus, Helsingborg, Skåne County
  - Sundsvalls hospital, Sundsvall, Västernorrland County
  - Sunderby Hospital, Luleå
  - Umea University Hospital, Umeå